CLINICAL TRIAL: NCT00216138
Title: A Single Arm Phase II Trial of Docetaxel and Capecitabine for the First Line Treatment of Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN): Hoosier Oncology Group HN02-40
Brief Title: Docetaxel and Capecitabine for First Line Treatment of Metastatic Squamous Cell Carcinoma of the Head & Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis results did not meet criteria for second stage of trial
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Sanofi (Industry); Hoffmann-La Roche (Industry); Walther Cancer Institute (Other)
Responsible Party: David Potter, M.D., Hoosier Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HOG HN02-40
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Capecitabine; Premedication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Docetaxel + Capecitabine
  Interventions: Drug: Docetaxel; Drug: Capecitabine; Drug: Premedication

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 60 mg/m2 for 60 minutes, day 1 of each cycle
Drug: Capecitabine — Capecitabine 825 mg/m2 po bid, days 1-14
Drug: Premedication — Dexamethasone and antiemetic premedication

SUMMARY:
Recent progress in treatment of recurrent/metastatic SCCHN has been made with the introduction of the taxanes. Docetaxel as a single agent has a response rate of 22-42% and 17% in patients with recurrent disease. Capecitabine is an oral fluoropyrimidine prodrug that is converted into 5-FU. Previous studies have shown that the capecitabine/docetaxel combination has a synergistic inhibition of tumor growth, resulting in significantly superior efficacy in time to disease progression (TTP), overall survival, median survival and objective tumor response rate compared to docetaxel alone.

This trial will investigate the efficacy the combination of docetaxel and capecitabine in treating patients with recurrent/metastatic SCCHN.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Dexamethasone and antiemetic premedication1.
* Docetaxel: 60 mg/m2 for a 60 minute infusion day 1 of each cycle
* Capecitabine: 825 mg/m2 po BID Days 1-14

Repeat every 21 days until tumor progression or toxicity that requires discontinuation of therapy

Performance status: ECOG performance status 0 or 1

Life expectancy: At least 3 months

Hematopoietic:

* ANC of > 1,500/mm3
* Platelets > 100,000/mm3
* Hemoglobin > 8 gm/dl

Hepatic:

* Total Bilirubin £ ULN
* Albumin > 3
* Maximum Alk Phos > 2.5 x < 5 x ULN

Renal:

* Creatinine clearance of > 50 ml/ min (by Cockcroft-Gault)

Cardiovascular:

* No decompensated congestive heart failure or active angina.
* Clinically significant cardiac disease not well controlled with medication (eg. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction in the past 12 months is not allowed.

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic squamous cell carcinoma of the head and neck.
* Recurrent/metastatic disease not amenable to surgery or salvage chemoradiation.
* Unidimensional measurable disease according to the RECIST
* In-field recurrence, within a prior radiation field only, distant metastatic disease
* Both in-field and metastatic sites of disease will require evaluation by a Radiation Oncologist to consider local radiation therapy first and will be eligible for possible enrollment one month after completion of the radiation therapy.
* Negative pregnancy test
* Patients may have received prior chemotherapy as part of chemoradiation or induction chemotherapy for initial treatment of disease confined to the head and neck region - Patients must have fully recovered from any prior radiation therapy

Exclusion Criteria:

* Patients who have relapsed < 6 months after completing a combined modality curative treatment that included a fluoropyrimidine or taxanes
* No brain metastases
* No major neurological disease, including stroke
* No prior chemotherapy regimen for recurrent/metastatic disease
* No prior history of capecitabine usage
* No prior history of docetaxel usage except in the induction setting for head and neck cancer which has been completed for greater than 6 months prior to beginning protocol therapy
* No past hypersensitivity to taxanes or 5 FU
* No hypersensitivity to docetaxel or other drugs formulated with polysorbate 80
* No current use of warfarin
* Patients must not be receiving ketoconazole, midazolam, erythromycin, orphenadrine, troleandomycin, cyclosporine or antiepileptics
* Patients must not be treated with any of the following on protocol therapy or within 28 days prior to beginning protocol therapy: sorivudine, brivudine, cimetidine, allopurinol
* Patients must have fully recovered from any prior surgery
* No known HIV seropositivity.
* No serious uncontrolled medical condition, uncontrolled peptic ulcer disease or malabsorption syndrome
* No peripheral neuropathy > grade 1
* Patients with a percutaneous gastrostomy (PEG) must be able take medications by tube.
* No daily consumption of alcohol
* No active infection
* No prior history of malignancy in the last 5 years, excluding in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin or Gleason Grade < VII organ confined prostate cancer.
* No current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
- To assess response rate in a group of patients receiving combination therapy with docetaxel and capecitabine | 24 months

SECONDARY OUTCOMES:
To assess toxicity of the combination | 24 months
To determine whether the status of calpain, calpain activation,(EGFR) expression, Cox-2 expression, TS, TP, DPD, and/or CYP3A4/CYP3A5 will predict treatment | 24 months
Efficacy and safety analyses on special sub-cohorts | 24 months
To determine the progression free survival and overall survival | 24 months
To assess change in analgesic usage with this protocol therapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Potter, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (18):
- United States (18):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - University of Chicago, Chicago, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Center for Hematology-Oncology of S Michigan, Jackson, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Methodist Cancer Center, Omaha, Nebraska

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/